CLINICAL TRIAL: NCT03093584
Title: Auricular Acupuncture (AA) vs. Expressive Writing in Treatment of Pre-exam Anxiety - Randomised Crossover Study in Medical Students
Brief Title: Auricular Stimulation vs. Expressive Writing for Exam Anxiety
Acronym: AA_EW_Anxi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BB 037/14
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auricular stimulation (Active Comparator): Auricular acupuncture with indwelling fixed auricular acupuncture needles
  Interventions: Device: Auricular acupuncture
- Expressive writing (Experimental): Expressive writing - sharing the emotional expectations in front of forthcoming exam
  Interventions: Behavioral: Expressive writing
- No intervention (No Intervention): No intervention, just observation and monitoring of outcome measures

INTERVENTIONS:
Device: Auricular acupuncture — Auricular acupuncture with indwelling fixed auricular acupuncture needles
  Arms: Auricular stimulation
Behavioral: Expressive writing — Expressive writing is a standard psychological method in treatment of exam anxiety
  Arms: Expressive writing

SUMMARY:
Title of the study: Auricular acupuncture (AA) vs. expressive writing for pre-exam anxiety - a randomised crossover study

Study period: 04 / 2014 - 07 / 2014

Principal Investigator: Prof. Dr. T. Usichenko Department of Anaesthesiology and Intensive Care Medicine University Medicine of Greifswald

Aim of the study: To investigate the anxiolytic effect of AA vs. expressive writing and vs. no intervention in students, passing the oral exams in anatomy at the University of Greifswald

Design: Prospective randomised crossover trial

Interventions: 1. AA using indwelling fixed needles, retained 24 h in situ 2. Expressive writing

Number of volunteers: N = 40

Healthy medical students at the University of Greifswald Participants of the anatomy exams in spring/summer 2014 Without previous anxiolytic, sedative and analgesic medication No pregnancy or lactating Informed consent

Outcome measures: Anxiety level Heart rate, blood pressure Salivary α-amylase

ELIGIBILITY:
Inclusion Criteria:

1. Medical students at the University of Greifswald
2. Going to take part in oral exams of human anatomy
3. Participants without previous anxiolytic medication
4. Ability to express the thoughts and emotions ("expressive writing")
5. Written informed consent

Exclusion Criteria:

1. Recidivist alcoholics
2. Local auricular skin infection
3. Pregnant or lactating women
4. Participants with prosthetic or damaged cardiac valves, intracardiac and intravascular shunts, hypertrophic cardiomyopathy and mitral valve prolaps (risk of bacterial endocarditis according to guidelines of AHA)
5. Participants who are unable to understand the consent form
6. History of psychiatric disease

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Intensity of anxiety | 2 days
  State-trait-Anxiety Inventory

SECONDARY OUTCOMES:
salivary alpha-amylase | 1 day
  enzymatic activity of salivary alpha-amylase
heart rate | 1 day
  heart rate
blood pressure | 1 day
  blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Taras Usichenko, MD. PhD, Principal Investigator — University Medicine of Greifswald

IPD SHARING:
Plan to Share IPD: Undecided